CLINICAL TRIAL: NCT02731508
Title: Bihemispheric Modulation of the Motor Cortex by Repetitive Transcranial Direct Current Stimulation After Stroke
Brief Title: Repetitive Bihemispheric Transcranial Direct Current Stimulation After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-03-003C
Record Dates: First submitted 2016-02-15; First posted 2016-04-07 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Stroke
Keywords: Transcranial Direct Current Stimulation; Neuroplasticity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- True stimulation (Experimental): True repetitive bihemispheric transcranial direct current stimulation, anodal at ipsilesional M1 while cathodal at contralesional M1, daily 20 minutes for 20 sessions
  Interventions: Device: Bihemispheric transcranial direct current stimulation
- Sham stimulation (Sham Comparator): Repetitive bihemispheric transcranial direct current stimulation, as the experimental stimulation condition but only for 120 seconds
  Interventions: Device: Bihemispheric transcranial direct current stimulation

INTERVENTIONS:
Device: Bihemispheric transcranial direct current stimulation — 5x5 cm tDCS electrode over C3 or C4 (10-20 system) with concurrent rehabilitation

SUMMARY:
Non-invasive repetitive bi-hemispheric transcranial direct current stimulation (tDCS) may restore post-stroke bi-hemispheric balance by increase peri-lesional cortex activity and suppress abnormal inhibition from non-lesional hemisphere, and therefore enhance after-effects of rehabilitation. In this double-blind, randomized controlled trial, investigators aim to investigate whether multi-session, bihemispheric tDCS to the primary motor cortex (M1) in combination with upper extremity rehabilitation therapy affected motor functional outcome, ipsilesional motor circuit excitability using transcranial magnetic stimulation (TMS) and magnetoencephalography (MEG) measures.

DETAILED DESCRIPTION:
Investigators will consecutively enroll subacute (2-6 weeks after stroke onset) patients with first-time, unilateral, ischemic subcortical stroke in the middle cerebral artery territory with mild to moderate hand weakness. All subjects will be randomly allocated to receive daily bihemispheric tDCS (anodal tDCS to ipsilesional M1 and cathodal tDCS to contralesional M1 with 2 mA stimulation for 20 min) or daily sham tDCS (same but stimulation for only 30 seconds) with simultaneous physical/occupational therapy, for total 10 sessions. Changes in upper extremity motor function score (Fugl-Meyer test and Action Research Arm test), corticospinal excitability from the transcranial magnetic stimulation(TMS), and sensorimotor oscillations from the magnetoencephalography (MEG) will be assessed before and after intervention, as well as 3 months after stroke. All stroke patients will receive tDCS and standard medical, rehabilitation treatments in rehabilitation ward.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years old
* Patients with first-time, unilateral, ischemic stroke with contralateral mild to moderate hand weakness
* Brain MRI confirmed subcortical stroke in the middle cerebral artery territory
* Post-stroke 2-6 weeks with stable clinical condition

Exclusion Criteria:

* Stroke with cortical lesions
* Containing metal implants (such as implanted electrodes, pacemakers)
* Sensitive or fear of electromagnetic waves
* Pregnant women
* History of alcohol or drug abuse
* History of seizures or epilepsy
* Claustrophobia
* Other significant disease or neuropsychiatric disorders

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-10; Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer test | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  stroke motor function scale

SECONDARY OUTCOMES:
Action Research Arm test | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  stroke motor function scale
Modified Rankin Scale | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  Global disability poststroke
Resting state functional connectivity | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  Functional MRI
Motor evoked potential | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  Transcranial magnetic stimulation test
Active motor threshold | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  Transcranial magnetic stimulation test
Ipsilateral silent period | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  Transcranial magnetic stimulation test
Short interval intracortical inhibition | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  Transcranial magnetic stimulation test
Motor task ERD peak amplitude | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  magnetoencephalography
Motor task ERS peak amplitude | baseline, change from baseline after 2 weeks' intervention, change from baseline at 3 months after stroke
  magnetoencephalography

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu SP, Lu CF, Lin BF, Tang CW, Kuo IJ, Tsai YA, Guo CY, Lee PL, Shyu KK, Niddam DM, Lee IH. Effects of bihemispheric transcranial direct current stimulation on motor recovery in subacute stroke patients: a double-blind, randomized sham-controlled trial. J Neuroeng Rehabil. 2023 Feb 27;20(1):27. doi: 10.1186/s12984-023-01153-4. PMID 36849990